CLINICAL TRIAL: NCT03699020
Title: Acceptance and Commitment Therapy to Address the Psychosocial Co-Morbidities of Chronic Pain in Aging People Living With HIV
Brief Title: Acceptance and Commitment Therapy for Aging People Living With HIV in Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Maile Young Karris, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 180837; 1R03AG060183-01 (NIH)
Record Dates: First submitted 2018-07-12; First posted 2018-10-09 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: HIV/AIDS; Chronic Pain
Keywords: HIV; Chronic Pain; Acceptance and Commitment Therapy; Behavioral Intervention; Older Adults
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Chronic Pain | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance and Commitment Therapy (ACT) (Experimental): The intervention will consists of eight weekly two hour group ACT sessions led by trained lay personnel and followed by homework. ACT is a behavioral therapy.
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT)
- Education Control (Experimental): Consists of eight weekly two hour group chronic pain education sessions led by trained lay personnel and followed by homework.
  Interventions: Other: Chronic Pain Education

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy (ACT) — Empirically based behavioral intervention that encourages acceptance of circumstances with commitment and behavioral change strategies to improve psychological flexibility.
  Arms: Acceptance and Commitment Therapy (ACT)
Other: Chronic Pain Education — Education materials about living with chronic pain developed by Weill Cornell Universitys Translational Research Institute for Pain in Later Life
  Arms: Education Control

SUMMARY:
Chronic pain impacts a large proportion of aging people living with HIV (aPLWH) and involves factors directly related to HIV (neurotoxicity) and psychosocial co-morbidities common in aPLWH (i.e. social isolation and loneliness). The investigators hypothesize that novel interventions that acknowledge these psychosocial co-morbidities may improve the efficacy of chronic pain management and minimize the use of potentially dangerous medications. This grant proposes to adapt and pilot a pain psychotherapy approach using group acceptance and commitment therapy (ACT) in aPLWH with chronic pain.

DETAILED DESCRIPTION:
Chronic pain affects a very high proportion of aging people living with HIV (aPLWH) and is thought to be related to both direct toxicity of HIV and antiretroviral therapy (ART) and by psychosocial factors that negatively affect pain (i.e. loneliness, HIV stigma). PLWH are also at increased risk for prescription opiate misuse. However as PLWH age, non-opiate medications used for pain can contribute to other negative outcomes such as falls, altered mental status and gastrointestinal bleeding. Thus there is a critical need for the development of novel interventions in the management of chronic pain in aPLWH that consider the psychological co-morbidities of aging with HIV and that can minimize the need for prescription medications. Acceptance and commitment therapy (ACT) has previously been evaluated in older persons with chronic pain and has demonstrated higher levels of satisfaction and efficacy when compared to cognitive behavioral therapy (CBT). ACT has never been evaluated in aPLWH for chronic pain, but has theoretical advantages over CBT for this population. Specifically several negatively modifying factors of CBT efficacy such as cognitive deficits are common in aPLWH.

The overarching objective of this study is to determine the acceptability and feasibility of an ACT intervention for the management of chronic pain adapted to aPLWH. To accomplish this objective the investigators will 1) train lay personnel to perform ACT to determine feasibility of this approach for future implementation, 2) conduct uncontrolled group ACT in aPLWH to generate participant feedback and questionnaire data to inform ACT adaption with the assistance of a steering commitee, and 3) conduct a pilot randomized controlled trial (RCT) evaluating the acceptability of adapted ACT compared to pain education. At completion of this grant the investigators expect to have successfully trained lay personnel to perform group ACT, adapted ACT from quantitative and qualitative data collected from an uncontrolled study of group ACT, and determined whether ACT is acceptable and feasible as an intervention in aPLWH. These expected outcomes may benefit other aging populations with chronic pain that are enriched for psychosocial co-morbidities such as persons who inject drugs, the socioeconomically disadvantaged, and racial or gender minorities. This proposal is aligned with the Office of AIDS Research High Priorities to better understand "HIV-associated comorbidities" which includes pain and to "Reduce Health Disparities in treatment outcomes of those living with HIV/AIDS" and with the National Pain Strategy to "expand investment ... in the development of safe and effective pain treatments."

ELIGIBILITY:
Inclusion Criteria:

* HIV seropositive
* Diagnosis of chronic non cancer pain
* English speaking
* Deemed appropriate for study by primary care provider
* Consents to participation

Exclusion Criteria:

* Cancer associated pain
* Unwillingness to participate in audio recorded sessions
* Enrollment in hospice
* Moderate to severe neurocognitive deficits (MOCA < 16)
* Currently undergoing other psychotherapy for chronic pain

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- AntiViral Research Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data including quantitative (questionnaires, baseline data) and qualitative (focus group) data will be stored in our secure database and made available to researchers upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available twelve months after study has ended and for five years.
Access Criteria: Contact PI and submission of brief proposal to minimize duplication of effort and ensure research questions are answerable using IPD available.

REFERENCES:
- [Background] Merlin JS, Cen L, Praestgaard A, Turner M, Obando A, Alpert C, Woolston S, Casarett D, Kostman J, Gross R, Frank I. Pain and physical and psychological symptoms in ambulatory HIV patients in the current treatment era. J Pain Symptom Manage. 2012 Mar;43(3):638-45. doi: 10.1016/j.jpainsymman.2011.04.019. Epub 2011 Nov 23. PMID 22115794
- [Background] Silverberg MJ, Gore ME, French AL, Gandhi M, Glesby MJ, Kovacs A, Wilson TE, Young MA, Gange SJ. Prevalence of clinical symptoms associated with highly active antiretroviral therapy in the Women's Interagency HIV Study. Clin Infect Dis. 2004 Sep 1;39(5):717-24. doi: 10.1086/423181. Epub 2004 Aug 16. PMID 15356788
- [Background] Cervia LD, McGowan JP, Weseley AJ. Clinical and demographic variables related to pain in HIV-infected individuals treated with effective, combination antiretroviral therapy (cART). Pain Med. 2010 Apr;11(4):498-503. doi: 10.1111/j.1526-4637.2010.00802.x. Epub 2010 Mar 4. PMID 20210870
- [Background] Heaton RK, Franklin DR, Ellis RJ, McCutchan JA, Letendre SL, Leblanc S, Corkran SH, Duarte NA, Clifford DB, Woods SP, Collier AC, Marra CM, Morgello S, Mindt MR, Taylor MJ, Marcotte TD, Atkinson JH, Wolfson T, Gelman BB, McArthur JC, Simpson DM, Abramson I, Gamst A, Fennema-Notestine C, Jernigan TL, Wong J, Grant I; CHARTER Group; HNRC Group. HIV-associated neurocognitive disorders before and during the era of combination antiretroviral therapy: differences in rates, nature, and predictors. J Neurovirol. 2011 Feb;17(1):3-16. doi: 10.1007/s13365-010-0006-1. Epub 2010 Dec 21. PMID 21174240
- [Background] Fishbain DA, Cutler R, Rosomoff HL, Rosomoff RS. Chronic pain-associated depression: antecedent or consequence of chronic pain? A review. Clin J Pain. 1997 Jun;13(2):116-37. doi: 10.1097/00002508-199706000-00006. PMID 9186019
- [Background] Lampe A, Doering S, Rumpold G, Solder E, Krismer M, Kantner-Rumplmair W, Schubert C, Sollner W. Chronic pain syndromes and their relation to childhood abuse and stressful life events. J Psychosom Res. 2003 Apr;54(4):361-7. doi: 10.1016/s0022-3999(02)00399-9. PMID 12670615
- [Background] Shippy RA, Karpiak SE. The aging HIV/AIDS population: fragile social networks. Aging Ment Health. 2005 May;9(3):246-54. doi: 10.1080/13607860412331336850. PMID 16019278
- [Background] Balderson BH, Grothaus L, Harrison RG, McCoy K, Mahoney C, Catz S. Chronic illness burden and quality of life in an aging HIV population. AIDS Care. 2013;25(4):451-8. doi: 10.1080/09540121.2012.712669. Epub 2012 Aug 15. PMID 22894702
- [Background] Moore RC, Moore DJ, Thompson WK, Vahia IV, Grant I, Jeste DV. A case-controlled study of successful aging in older HIV-infected adults. J Clin Psychiatry. 2013 May;74(5):e417-23. doi: 10.4088/JCP.12m08100. PMID 23759460
- [Background] Merlin JS, Westfall AO, Raper JL, Zinski A, Norton WE, Willig JH, Gross R, Ritchie CS, Saag MS, Mugavero MJ. Pain, mood, and substance abuse in HIV: implications for clinic visit utilization, antiretroviral therapy adherence, and virologic failure. J Acquir Immune Defic Syndr. 2012 Oct 1;61(2):164-70. doi: 10.1097/QAI.0b013e3182662215. PMID 22766967
- [Background] Vijayaraghavan M, Freitas D, Bangsberg DR, Miaskowski C, Kushel MB. Non-medical use of non-opioid psychotherapeutic medications in a community-based cohort of HIV-infected indigent adults. Drug Alcohol Depend. 2014 Oct 1;143:263-7. doi: 10.1016/j.drugalcdep.2014.06.044. Epub 2014 Jul 27. PMID 25107312
- [Background] Green TC, McGowan SK, Yokell MA, Pouget ER, Rich JD. HIV infection and risk of overdose: a systematic review and meta-analysis. AIDS. 2012 Feb 20;26(4):403-17. doi: 10.1097/QAD.0b013e32834f19b6. PMID 22112599
- [Background] Merlin JS, Zinski A, Norton WE, Ritchie CS, Saag MS, Mugavero MJ, Treisman G, Hooten WM. A conceptual framework for understanding chronic pain in patients with HIV. Pain Pract. 2014 Mar;14(3):207-16. doi: 10.1111/papr.12052. Epub 2013 Apr 1. PMID 23551857
- [Background] By the American Geriatrics Society 2015 Beers Criteria Update Expert Panel. American Geriatrics Society 2015 Updated Beers Criteria for Potentially Inappropriate Medication Use in Older Adults. J Am Geriatr Soc. 2015 Nov;63(11):2227-46. doi: 10.1111/jgs.13702. Epub 2015 Oct 8. PMID 26446832
- [Background] Keefe FJ, Kashikar-Zuck S, Opiteck J, Hage E, Dalrymple L, Blumenthal JA. Pain in arthritis and musculoskeletal disorders: the role of coping skills training and exercise interventions. J Orthop Sports Phys Ther. 1996 Oct;24(4):279-90. doi: 10.2519/jospt.1996.24.4.279. PMID 8892142
- [Background] Sotsky SM, Glass DR, Shea MT, Pilkonis PA, Collins JF, Elkin I, Watkins JT, Imber SD, Leber WR, Moyer J, et al. Patient predictors of response to psychotherapy and pharmacotherapy: findings in the NIMH Treatment of Depression Collaborative Research Program. Am J Psychiatry. 1991 Aug;148(8):997-1008. doi: 10.1176/ajp.148.8.997. PMID 1853989
- [Background] McCracken LM, Morley S. The psychological flexibility model: a basis for integration and progress in psychological approaches to chronic pain management. J Pain. 2014 Mar;15(3):221-34. doi: 10.1016/j.jpain.2013.10.014. PMID 24581630
- [Background] McCracken LM, Vowles KE. Acceptance and commitment therapy and mindfulness for chronic pain: model, process, and progress. Am Psychol. 2014 Feb-Mar;69(2):178-87. doi: 10.1037/a0035623. PMID 24547803
- [Background] Hofmann SG, Asmundson GJG. Acceptance and mindfulness-based therapy: new wave or old hat? Clin Psychol Rev. 2008 Jan;28(1):1-16. doi: 10.1016/j.cpr.2007.09.003. Epub 2007 Sep 18. PMID 17904260
- [Background] Prevedini AB, Presti G, Rabitti E, Miselli G, Moderato P. Acceptance and commitment therapy (ACT): the foundation of the therapeutic model and an overview of its contribution to the treatment of patients with chronic physical diseases. G Ital Med Lav Ergon. 2011 Jan-Mar;33(1 Suppl A):A53-63. PMID 21488484
- [Background] Alonso-Fernandez M, Lopez-Lopez A, Losada A, Gonzalez JL, Wetherell JL. Acceptance and Commitment Therapy and Selective Optimization with Compensation for Institutionalized Older People with Chronic Pain. Pain Med. 2016 Feb;17(2):264-77. doi: 10.1111/pme.12885. PMID 26304771
- [Background] Wetherell JL, Petkus AJ, Alonso-Fernandez M, Bower ES, Steiner AR, Afari N. Age moderates response to acceptance and commitment therapy vs. cognitive behavioral therapy for chronic pain. Int J Geriatr Psychiatry. 2016 Mar;31(3):302-8. doi: 10.1002/gps.4330. Epub 2015 Jul 28. PMID 26216753
- [Background] Petkus AJ, M A, Wetherell JL. Acceptance and Commitment Therapy with Older Adults: Rationale and Considerations. Cogn Behav Pract. 2013 Feb;20(1):47-56. doi: 10.1016/j.cbpra.2011.07.004. PMID 26997859
- [Background] Moitra E, Herbert JD, Forman EM. Acceptance-based behavior therapy to promote HIV medication adherence. AIDS Care. 2011 Dec;23(12):1660-7. doi: 10.1080/09540121.2011.579945. Epub 2011 Jul 7. PMID 21732897
- [Background] Chen EK, Reid MC, Parker SJ, Pillemer K. Tailoring evidence-based interventions for new populations: a method for program adaptation through community engagement. Eval Health Prof. 2013 Mar;36(1):73-92. doi: 10.1177/0163278712442536. Epub 2012 Apr 19. PMID 22523308
- [Background] McGrath PJ, Walco GA, Turk DC, Dworkin RH, Brown MT, Davidson K, Eccleston C, Finley GA, Goldschneider K, Haverkos L, Hertz SH, Ljungman G, Palermo T, Rappaport BA, Rhodes T, Schechter N, Scott J, Sethna N, Svensson OK, Stinson J, von Baeyer CL, Walker L, Weisman S, White RE, Zajicek A, Zeltzer L; PedIMMPACT. Core outcome domains and measures for pediatric acute and chronic/recurrent pain clinical trials: PedIMMPACT recommendations. J Pain. 2008 Sep;9(9):771-83. doi: 10.1016/j.jpain.2008.04.007. Epub 2008 Jun 17. PMID 18562251

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants were randomized to groups shortly after enrollment.
Period: Overall Study
Arm/Group | Acceptance and Commitment Therapy (ACT) | Education Control
Started | 7 | 5
Intervention Attendance Completion | 4 | 3
Completed | 4 | 3
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Population: These participants were randomized, however once the intervention or control started several participants opted to no longer continue
Groups:
- Total: Total of all reporting groups
Arm/Group | Acceptance and Commitment Therapy (ACT) | Education Control | Total
Number analyzed (Participants) | 7 | 5 | 12
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58 [57.5 to 66.5] | 57 [57 to 62] | 58 [57 to 62.25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 6 | 3 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 4 | 4 | 8
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 5 | 12
Years living with HIV [Median (Inter-Quartile Range); unit: years] — Years participant has been living with HIV. Participant reported, at least from date of diagnosis
  years | 24 [22.5 to 24] | 29 [27 to 33] | 24 [23 to 27.5]
Years on antiretroviral therapy [Median (Inter-Quartile Range); unit: years] — Years that participant has been taking antiretroviral therapy for HIV
  years | 24 [22.5 to 24] | 23 [14 to 24] | 23 [19.3 to 24.5]
Current HIV Viral Load [Median (Inter-Quartile Range); unit: HIV copies/mL] — Viral load is measured in blood and represented as "x" copies/mL. Of note we used "0" for undetectable or < 20 copies/mL
  HIV copies/mL | 0 [0 to 0] | 46 [46 to 184] | 46 [46 to 88]
Current CD4 T cell count [Median (Inter-Quartile Range); unit: cells/m3] — CD4+ T cells, total number of cells per m3
  cells/m3 | 716 [639 to 1007] | 1051 [408 to 1161] | 1051 [513.8 to 1053.3]
Veterans Aging Cohort Study Index [Median (Inter-Quartile Range); unit: units on a scale] — The VACS 1.0 Index characterize the 5 year mortality risk in people with HIV. This Index incorporates age, CD4 T cell count, HIV-1 RNA, hemoglobin, Fib-4 index, eGRF, and Hepatitis C coinfection to create a total score (score range 0 to 164). A score of 0 equates to 1.8% predicted all cause 5-year mortality; a 164 has >85.8% predicted all cause 5-year mortality. This means the higher the VACS index the higher the probability of 5-year mortality due to all causes.
  units on a scale | 33 [28 to 34] | 27 [12 to 39] | 27 [15.8 to 37.8]
Total # pain medications [Median (Inter-Quartile Range); unit: number of medications] — We added unique medications (prescribed and over the counter) that participants stated they used daily for pain management including opioids, muscle relaxants, medications for neuropathy, NSAIDS, acetaminophen etc.
  number of medications | 2 [0 to 3] | 2 [0 to 3] | 2 [0 to 3]
Total # of opioid/opiates prescribed [Median (Inter-Quartile Range); unit: total # of opioid/opiates prescribed] — Total number of unique prescribed opioid/opiates participants were taking. We did not calculate morphine miligram equivalents.
  total # of opioid/opiates prescribed | 0 [0 to 0.25] | 0.5 [0.25 to 0.75] | 0.5 [0 to 0.75]
Baseline CPAQ-R Activity Engagement [Median (Inter-Quartile Range); unit: units on a scale] — The 20 item Chronic Pain Acceptance Questionnaire-Revised measures acceptance of pain. There are two factors 1) activity engagement (pursuit of life activities regardless of pain) and 2) pain willingness (the recognition that avoidance and control are often unworkable methods of adapting to chronic pain). Higher scores indicate higher levels of acceptance
  The activity engagement scale has 11 items each rated from 0 (never true) to 6 (always true). Scores are added and the range of the activity engagement scale is 0 (no acceptance of pain) to 66 (high acceptance of pain).
  units on a scale | 42 [37 to 53] | 25.5 [21.8 to 28.8] | 34 [27 to 47]
Baseline CPAQ-R Pain Willingness [Median (Inter-Quartile Range); unit: units on a scale] — The 20 item Chronic Pain Acceptance Questionnaire-Revised measures acceptance of pain in regards to 1) activity engagement (pursuit of life activities regardless of pain) and 2) pain willingness (the recognition that avoidance and control are often unworkable methods of adapting to chronic pain). Higher scores indicate higher levels of acceptance
  The pain willingness scale includes 9 items and all items are rated from 0 (never true) to 6 (always true). Scores are added and the range is 0 (no acceptance of pain) to 54 (high acceptance of pain).
  units on a scale | 32 [20.5 to 40.5] | 32 [31.3 to 33.5] | 32 [26.5 to 39]
Baseline CPAQ-R (revised) Total Score [Median (Inter-Quartile Range); unit: units on a scale] — The 20 item Chronic Pain Acceptance Questionnaire-Revised (CPAQ-R) is designed to measure acceptance of pain. There are two factors identified 1) Activity engagement (pursuit of life activities regardless of pain) and 2) pain willingness (the recognition that avoidance and control are often unworkable methods of adapting to chronic pain). Higher scores indicate higher levels of acceptance. Range is 0 (no acceptance) to 120 (high acceptance)
  units on a scale | 68 [66 to 76] | 56 [55.3 to 58.5] | 66 [60.5 to 69.5]
Brief Pain Inventory: Pain Severity (worse) [Median (Inter-Quartile Range); unit: units on a scale] — Brief Pain Inventory (BPI) short form measures two domains 1) pain intensity (severity) and 2) the impact of pain on functioning (interference). The BPI does not have a scoring algorithm. Most researcher use ratings of "worse" and "average" pain scores to describe pain intensity. The range is from 0 (no pain) to 10 (pain as bad as you can imagine.
  units on a scale | 8 [7.5 to 9.5] | 6 [5.75 to 6.5] | 8 [6.5 to 8.5]
Brief Pain Inventory: Pain Severity (average) [Median (Inter-Quartile Range); unit: units on a scale] — Brief Pain Inventory (BPI) short form measures two domains 1) pain intensity (severity) and 2) the impact of pain on functioning (interference). The BPI does not have a scoring algorithm. Most researcher use ratings of "worse" and "average" pain scores to describe pain intensity. The range is from 0 (no pain) to 10 (pain as bad as you can imagine.
  units on a scale | 8 [8 to 9] | 4.5 [3.25 to 5.5] | 8 [6 to 8]
Brief Pain Inventory: Pain interference [Median (Inter-Quartile Range); unit: units on a scale] — Brief Pain Inventory short form also measures the impact of pain on functioning (interference). Seven questions inquire about the how much pain interferes with general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Each of these areas are scored from 0 (does not interfere) to 10 (completely interferes). Pain interference is reported as a mean of these 7 unique areas.
  units on a scale | 5 [4 to 7.5] | 5 [4.1 to 5.8] | 5 [4 to 6.8]
Pain Knowledge Test % Correct [Median (Inter-Quartile Range); unit: % questions answered correctly] — To evaluate the impact or not of the control (pain education) a general pain knowledge test was provided to all participants. We then provide the median of the % of questions that participants answered correctly on the test.
  % questions answered correctly | 80 [70 to 85] | 75 [67.5 to 82.5] | 80 [70 to 85]

OUTCOME MEASURES:

1. Primary Outcome: Change in Chronic Pain Acceptance Questionnaire (CPAQ) Week 0 to Week 6
Description: Change in Chronic Pain Acceptance Questionnaire or CPAQ from study entry to end of intervention. This scale measures acceptance of chronic pain and measures two factors: activity engagement (pursuit of life activities regardless of pain) and pain willingness (recognition that avoidance and control are often unworkable methods of adapting to chronic pain). A total of 20 items represents these two factors and the items are rated on a 7-point scale from 0 (never true) to 6 (always true). Scoring the CPAQ requires adding the summed items for activity engagement and pain willingness for a total score. Thus the range of scores is from 0 (no acceptance) to 120 (full acceptance). Change in scale will be represented by the difference in CPAQ total score from baseline to week 6.
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Acceptance and Commitment Therapy (ACT): The intervention will consists of six weekly two hour group ACT sessions led by trained lay personnel and followed by homework. ACT is a behavioral therapy.
  Acceptance and Commitment Therapy (ACT): Empirically based behavioral intervention that encourages acceptance of circumstances with commitment and behavioral change strategies to improve psychological flexibility.
- Education Control: Consists of six weekly two hour group chronic pain education sessions led by trained lay personnel and followed by homework.
  Chronic Pain Education: Education materials about living with chronic pain developed by Weill Cornell Universitys Translational Research Institute for Pain in Later Life
Arm/Group | Acceptance and Commitment Therapy (ACT) | Education Control
Number analyzed (Participants) | 4 | 3
score on a scale | 5 [2.5 to 7] | 13 [6 to 29]

2. Secondary Outcome: Change in Chronic Pain Acceptance Questionnaire Week 0 to Week 3
Description: Change in Chronic Pain Acceptance Questionnaire or CPAQ from study entry to end of intervention. This scale measures acceptance of chronic pain and measures two factors: activity engagement (pursuit of life activities regardless of pain) and pain willingness (recognition that avoidance and control are often unworkable methods of adapting to chronic pain). A total of 20 items represents these two factors and the items are rated on a 7-point scale from 0 (never true) to 6 (always true). Scoring the CPAQ requires adding the summed items for activity engagement and pain willingness for a total score. Thus the range of scores is from 0 (no acceptance) to 120 (full acceptance). Change in scale will be represented by the difference in CPAQ total score from baseline to week 3.
Time Frame: 3 weeks
Measure: Median (Inter-Quartile Range); unit: change in score from 0 to 6 weeks.
Arm/Group | Acceptance and Commitment Therapy (ACT) | Education Control
Number analyzed (Participants) | 4 | 3
change in score from 0 to 6 weeks. | 5.5 [4.75 to 6.25] | 13 [5 to 21]

3. Secondary Outcome: Brief Pain Inventory Interference Subscale
Description: Change in the Brief Pain Inventory (BPI) Interference subscale from week 0 to 6. The BPI allows persons to rate the severity of their pain (pain severity subscale) and the degree to which their pain interferes with feeling and function (interference subscale). The severity scale assess pain at its "worst, least, average and now". These 4 items are ranked from 0 (no pain) to 10 (pain as bad as you can imagine). Most commonly single items of "worst" and "average" are used to represent severity. A composite of the four items (mean severity score) is often also presented. Pain interference has 7 items "general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life" and is scored from 0 (does not interfere) to 10 (completely interferes). Pain interference subscale is scored as the mean of the seven interference items. Change in BPI interference subscale will be represented by the difference in mean interference from baseline to week 6.
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Acceptance and Commitment Therapy (ACT) | Education Control
Number analyzed (Participants) | 4 | 3
score on a scale | -1.71 [-2.57 to -0.86] | -0.14 [-1.21 to 0.21]

4. Secondary Outcome: Change in Pain Education Score
Description: Difference from Week 0 to 6 in proportion of pain knowledge questions answered correctly.
Time Frame: Week 0 to Week 6
Measure: Median (Inter-Quartile Range); unit: proportion of correct answers
Arm/Group | Acceptance and Commitment Therapy (ACT) | Education Control
Number analyzed (Participants) | 4 | 3
proportion of correct answers | 0.05 [-0.075 to 0.175] | 0.1 [0.1 to 0.2]

ADVERSE EVENTS:
Time Frame: 2 years
Description: Adverse events would be defined as events reported by participants and study staff
Arm/Group | Acceptance and Commitment Therapy (ACT) | Education Control
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3

LIMITATIONS AND CAVEATS:
We hypothesize our ability to recruit and engage participants was impaired by the COVID-19 pandemic. Barriers included halting of non-covid studies, IRB approval for remote delivery of the intervention, disinterest in research participation in the context of COVID, lack of access to reliable internet connectivity and unfamiliarity with video visits.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-22): https://cdn.clinicaltrials.gov/large-docs/20/NCT03699020/Prot_SAP_000.pdf